CLINICAL TRIAL: NCT03124043
Title: Get In Touch Phase 2 - Evaluating a Diabetes Care Support Program Facilitated by Cellular-enabled Glucose Meters, a Randomized Crossover Trial
Brief Title: Get In Touch Phase 2
Acronym: GIT-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Livongo Health (Industry)
Responsible Party: Principal Investigator, Daniel Amante, Program Director, University of Massachusetts, Worcester
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: H00005902
Record Dates: First submitted 2016-12-19; First posted 2017-04-21 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention First (Experimental): Participants in Intervention First were enrolled in the intervention for the first 6 months of study participation followed by a return to usual care for the following 6 months. The intervention included provision of a cellular-enable glucose meter and enrollment in the Livongo for Diabetes support program that provided both in-the-moment and scheduled support, both provided by Livongo Health Inc.
  Interventions: Other: Livongo for Diabetes program
- Intervention Second (Experimental): Participants in the 'Intervention Second" received usual care for the first 6 months of study participation followed by enrollment in the intervention for the following 6 months. The intervention included provision of a cellular-enable glucose meter and enrollment in the Livongo for Diabetes support program that provided both in-the-moment and scheduled support, both provided by Livongo Health Inc.
  Interventions: Other: Livongo for Diabetes program

INTERVENTIONS:
Other: Livongo for Diabetes program — See description in arm/group description.

SUMMARY:
The objective of the Get In Touch - Phase 2 (GIT-2) study was to evaluate a diabetes care support intervention facilitated by cellular-enabled glucose meters in adults with persistent poor control of type 2 diabetes.

DETAILED DESCRIPTION:
A 2-group randomized crossover trial comparing usual care to a diabetes care support intervention among patients with repeated HbA1c recordings greater than 8.0 percent during the previous 12 months. The intervention included 6 months of enrollment in Livongo for Diabetes, a Certified Diabetes Educator (CDE) based remote diabetes monitoring program facilitated by cellular-enabled glucose meters, with additional remote monitoring by their usual care team. HbA1c levels were recorded at enrollment and 3, 6, 9, and 12 months post enrollment. Questionnaire data were collected at baseline, 6 months, and 12 months post enrollment. Primary outcomes evaluated were change in HbA1c and treatment satisfaction at the 6 month endpoint with secondary outcomes of change in HbA1c and treatment satisfaction at the 12 month endpoint.

ELIGIBILITY:
Inclusion Criteria:

* speak English, having type 2 diabetes with two consecutive HbA1c recordings greater than 8.0% over the previous 12 months at the time of recruitment

Exclusion Criteria:

* excluded if they were cognitively impaired, pregnant, or prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-04; Primary Completion 2016-09 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | During 6-month enrollment in Intervention
  The primary physiological outcome of this study was change in HbA1c during enrollment in the intervention compared to change while receiving usual care.

SECONDARY OUTCOMES:
Change in Treatment Satisfaction | During 6-month enrollment in intervention
  The secondary outcome of this study was change in treatment satisfaction during enrollment in the intervention compared to change while receiving usual care. Treatment Satisfaction Change was measured using the Diabetes Treatment Satisfaction Questionnaire Change (DTSQc) scale.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Thompson, MD, Principal Investigator — UMass Medical School

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Amante DJ, Harlan DM, Lemon SC, McManus DD, Olaitan OO, Pagoto SL, Gerber BS, Thompson MJ. Evaluation of a Diabetes Remote Monitoring Program Facilitated by Connected Glucose Meters for Patients With Poorly Controlled Type 2 Diabetes: Randomized Crossover Trial. JMIR Diabetes. 2021 Mar 11;6(1):e25574. doi: 10.2196/25574. PMID 33704077